CLINICAL TRIAL: NCT02202356
Title: A Randomized, Double-blind, Placebo-controlled, 2-Part Study of Orally Administered ALS-008176 to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Dosing and Multiple Ascending Dosing in Infants Hospitalized With Respiratory Syncytial Virus (RSV) Infection
Brief Title: A Study of ALS-008176 in Infants Hospitalized With RSV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alios Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALS-8176-503; 2013-005104-33 (EudraCT Number)
Record Dates: First submitted 2014-07-23; First posted 2014-07-29 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — 4'-chloromethyl-2'-deoxy-3',5'-di-O-isobutyryl-2'-fluorocytidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (4):
- ALS-008176 Single Dose (Experimental): Single dose of ALS-008176 administered orally as a suspension
  Interventions: Drug: ALS-008176
- Placebo Single Dose (Placebo Comparator): Single dose of placebo administered orally as a suspension
  Interventions: Drug: Placebo
- ALS-008176 Multiple Doses (Experimental): Multiple doses of ALS-008176 administered orally as a suspension
  Interventions: Drug: ALS-008176
- Placebo Multiple Doses (Placebo Comparator): Multiple doses of placebo administered orally as a suspension
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALS-008176
  Arms: ALS-008176 Multiple Doses; ALS-008176 Single Dose
Drug: Placebo
  Arms: Placebo Multiple Doses; Placebo Single Dose

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK) and anti-viral effect of single and multiple doses of ALS-008176 in infants hospitalized with respiratory syncytial virus (RSV)

ELIGIBILITY:
Inclusion Criteria:

* Male or female infant who is ≥1.0 to ≤12.0 months of age (inclusive), defined at the time of hospital admission, or <28 days of age (neonate cohort only). Note: all subjects, including neonates, must have been discharged from the hospital after birth and are now being admitted due to an RSV related illness

Exclusion Criteria:

* Prematurity
* Receiving invasive endotracheal mechanical ventilation
* Poorly functioning gastrointestinal tract
* Anticipated to be discharged from the hospital in <24 hours from the time of randomization
* Prior exposure to palivizumab

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Baseline through 6 days post-dose
Physical Examinations | Baseline through 6 days post-dose
Vital Signs | Baseline through 6 days post-dose
12-Lead ECGs | Baseline through 6 days post-dose
Clinical Laboratory Results | Baseline through 6 days post-dose

SECONDARY OUTCOMES:
RSV viral RNA concentrations in nasal aspirates | Baseline through 6 days post-dose
Emergence of resistance | Baseline through 6 days post-dose
  Changes in RSV polymerase that result in reduced sensitivity to study drug
Pharmacokinetic parameters, including maximum and minimum drug concentrations | Baseline through 6 days post-dose
Pharmacokinetic parameters, including time to maximum concentration and half-life | Baseline through 6 days post-dose
Pharmacokinetic parameters, including area under concentration-time curves (AUCs) | Baseline through 6 days post-dose
Pharmacokinetic parameters, including apparent oral clearance (CL/F) and apparent volume of distribution at steady state (VDss/F) | Baseline through 6 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McClure, M.D., Study Director — Alios BioPharma
Locations (77):
- United States (17):
  - Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital Research Institute, Little Rock, Arkansas
  - Long Beach Memorial Medical Center/Miller Children's and Women's Hospital of Long Beach, Long Beach, California
  - Children's Hospital of Orange County, Orange, California
  - The University of California at San Diego, San Diego, California
  - LSU Health Sciences Center, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Children's Mercy, Kansas City, Missouri
  - University of Rochester, Rochester, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - The Research Institute at Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital/University of Tennessee, Memphis, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital/Baylor College of Medicine, Houston, Texas
  - The University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (5):
  - The Canberra Hospital, Canberra
  - Monash Medical Center, Melbourne
  - Women's and Children's Hospital, North Adelaide
  - The Royal Children's Hospital Melbourne, Parkville
  - Princess Margaret Hospital, Perth
- Canada (4):
  - The Children's Hospital Research Institute of Manitoba, Winnipeg, Manitoba
  - Canadian Centre for Vaccinology IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Chile (3):
  - Hospital Dr. Exequiel Gonzalez Cortes, San Miguel, Santiago Metropolitan
  - Complejo Asistencial Dr Sotero del Rio, Santiago
  - Hospital Padre Hurtado, Santiago
- Colombia (2):
  - Fundacion Cardio Infantil Instituto de Cardiologia, Bogotá
  - Hospital Pablo Tobon Uribe, Medellín
- France (2):
  - CHU Pellegrin / Pneumologie pediatrique, Bordeaux
  - Hopital Necker, Paris
- Japan (17):
  - Hirosaki National Hospital, Hirosaki-shi, Aomori
  - Chiba Children's Hospital, Chiba, Chiba
  - Ota Memorial Hospital, Ōta, Gunma
  - Gunma Children's Medical Center, Shibukawa-shi, Gunma
  - NHO Fukuyama Medical Center, Fukuyama, Hiroshima
  - Hokkaido P.W.F.A.C. Asahikawa-Kosei General Hospital, Asahikawa-shi, Hokkaido
  - NHO Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - NHO Shikoku Medical Center for Children and Adults, Takamatsu, Kagawa-ken
  - Okinawa Chubu Hospital, Urumi, Okinawa
  - Nakano Children's Hospital, Osaka, Osaka
  - National Hospital Organization Saitama National Hospital, Wako, Saitama
  - Tokyo Metropolitan Children's Medical Center, Fuchu-shi, Tokyo
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
  - Fukuoka Children's Hospital, Fukuoka
  - NHO Fukuoka Hospital, Fukuoka
  - Kochi Health Sciences Center, Kochi
  - Saitama Children's Medical Center, Saitama
- New Zealand (3):
  - Christchurch Clinical Study Trust, Christchurch
  - Hawke's Bay Hospital, Hastings
  - Wellington Hospital, Wellington
- Panama (3):
  - Hospital Materno Infantil Jose Dominog de Obaldila, David, Chiriquí Province
  - Hospital de Especialidades Pediatricas "Omar Torrijos Herrera", Panama City
  - Hospital del Nino, Panama City
- Institute for Mother and Child Care "Alfred Rusescu", Bucharest, Romania
- South Africa (3):
  - 2 Military Hospital, Cape Town
  - Kingsbury Hospital, Cape Town
  - Tygerberg Academic Hospital, Cape Town
- Taiwan (2):
  - Linkou Chang Gung Medical Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
- Thailand (4):
  - Chulalongkorn University Department of Pediatrics, Bangkok
  - Phramongkutklao Hospital Department of Pediatrics, Bangkok
  - Siriraj Hospital, Mahidol University Department of Pediatrics, Bangkok
  - Khon Kaen University Department of Pediatrics, Khon Kaen
- United Kingdom (11):
  - Bristol Royal Hospital for Children, Bristol, England
  - Alder Hey Children's Hospital, Liverpool, England
  - St. George's University of London, London, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, England
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Children's Hospital of Wales, Cardiff, Wales
  - Birmingham Children's Hospital, Birmingham
  - Royal Alexandra Children's Hospital, Brighton
  - Royal Manchester Children's Hospital, Manchester
  - Queens Medical Center, Nottingham
  - University of Oxford, Oxford

REFERENCES:
- [Derived] Oey A, McClure M, Symons JA, Chanda S, Fry J, Smith PF, Luciani K, Fayon M, Chokephaibulkit K, Uppala R, Bernatoniene J, Furuno K, Stanley T, Huntjens D, Witek J; 503 and RSV2004 Study Groups. Lumicitabine, an orally administered nucleoside analog, in infants hospitalized with respiratory syncytial virus (RSV) infection: Safety, efficacy, and pharmacokinetic results. PLoS One. 2023 Jul 19;18(7):e0288271. doi: 10.1371/journal.pone.0288271. eCollection 2023. PMID 37467213